CLINICAL TRIAL: NCT02120794
Title: Multi-Center, Prospective, Observational Study of the TS (Threshold Suspend) Feature With a Sensor-Augmented Pump System in Pediatric Patients With Type 1 Diabetes
Brief Title: Threshold Suspend in Pediatrics at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP287
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Pediatric; Threshold Suspend; Sensor augmented pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: single group
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 530G insulin pump (Experimental): Subjects will use 530G insulin pump with Threshold Suspend (TS) feature for one year.
  Interventions: Device: 530G Insulin pump

INTERVENTIONS:
Device: 530G Insulin pump — Subjects will use 530G insulin pump with Threshold Suspend (TS) feature for one year.

SUMMARY:
The study objective is to demonstrate that home use of Threshold Suspend (TS) is not associated with glycemic deterioration in pediatric patients with type 1 diabetes, as measured by change in A1C.

DETAILED DESCRIPTION:
This study is a longitudinal, multi-center trial that aims to observe the Threshold Suspend (TS) feature with a sensor-augmented insulin pump in patients 7-15 years with Type 1 diabetes. The study will measure the change in A1C from baseline over a period of one year while subjects are wearing the study pump.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 2 to 15 at time of screening
2. Subject has been diagnosed with type 1 diabetes mellitus and must have been diagnosed for at least one year prior to screening
3. Subject is currently transitioning from pump therapy, with or without continued glucose monitoring (CGM), to the 530G insulin pump system.
4. Subject is willing to perform greater than or equal to 4 finger stick blood glucose measurements daily
5. Subject is willing to perform required sensor calibrations
6. Subject is willing to wear the system (Pump, glucose sensors, meter) continuously throughout the study
7. Subject is willing to upload data every 21 days from the study pump
8. Subject must have Internet access and access to a computer system that meets the requirements for uploading the pumps. This may include use of family or friend's computer system with Internet access.
9. Subject is using either Humalog or Novolog at time of Screening and plans to use either of those insulins throughout the study

Exclusion Criteria:

1. Subject is actively participating in an investigational study (drug or device) wherein he/she is receiving treatment from an investigational study drug or investigational study device.
2. Women of child-bearing potential who have a positive pregnancy test at screening or plan to become pregnant during the course of the study
3. Subject is being treated for hyperthyroidism at time of screening
4. Subject has an abnormality (>1.8mg/dL) in creatinine at time of screening visit
5. Subject has an abnormality (out of reference range) in thyroid-stimulating hormone (TSH) at time of screening visit; If TSH is out of range, Free T3 and Free T4 will be tested; subject may be included with TSH out of range as long as Free T3 and Free T4 are in normal reference range.
6. Subject has taken any oral, injectable, or IV steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study
7. Subject is currently abusing illicit drugs
8. Subject is currently abusing prescription drugs
9. Subject is currently abusing alcohol
10. Subject is using pramlintide (Symlin) at time of screening
11. Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
12. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
13. Subject diagnosed with current eating disorder such as anorexia or bulimia
14. Subject has been diagnosed with chronic kidney disease that results in chronic anemia
15. Subject is on dialysis
16. Subject is already on a 530G system with CGM for 8 days or more.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2014-06; Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lee, M.D., Study Director — Medtronic Diabetes
Locations (16):
- United States (16):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Institute for Medical Research Excellence in Diabetes and Endocrinology, Sacramento, California
  - Madison Clinic for Pediatric Diabetes at UCSF, San Francisco, California
  - Stanford University, Stanford, California
  - SoCal Diabetes, Torrance, California
  - University of Colorado Health Science Center, Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Health System, Jacksonville, Florida
  - Park Nicollet Clinic - International Diabetes Center, Minneapolis, Minnesota
  - University of Minnesota Pediatric Endocrinology Clinic, Minneapolis, Minnesota
  - Children's Hospital and Clinics of Minnesota, Saint Paul, Minnesota
  - The Pediatric and Endocrine Diabetes Specialists, Las Vegas, Nevada
  - Stony Brook Children's Hospital, East Setauket, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children Hospital/Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 530G Insulin Pump
Started | 194
Completed | 136
Not Completed | 58
Not completed — Withdrawal by Subject | 43
Not completed — Adverse Event | 10
Not completed — Physician Decision | 4
Not completed — Due to insurance coverage | 1

BASELINE CHARACTERISTICS:
Arm/Group | 530G Insulin Pump
Number analyzed (Participants) | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 164
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: particpants]
  United States | 194

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change in A1C
Description: The overall mean change in A1C from baseline to 1 year will be estimated and compared by a non-inferiority test with an A1C margin of 0.4% and a significance level of 0.025 (one-sided). Among the 136 subjects who completed the study, 132 had both baseline and end of study A1c. Therefore, primary endpoint was based on 132 subjects.
Time Frame: Baseline and 1 year after screening
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | 530G Insulin Pump
Number analyzed (Participants) | 132
percentage | 0.26 [0.125 to 0.395]
Statistical Analysis 1: Comparison: 530G Insulin Pump; Test type: Non-Inferiority — non-inferiority test with an A1C margin of 0.4% and a significance level of 0.025 (one-sided); Mean Difference (Net) = 0.26, 95% CI 2-sided [0.125 to 0.395]

2. Secondary Outcome: Mean Change in A1C From Baseline to 1 Year, Stratified by Different A1c Subgroups
Description: Mean change in A1C from baseline to 1 year, stratified by different A1c subgroups: A1c below 7%. Among the 132 subjects with both baseline and end of study A1c, 3 had A1c below 7%
Time Frame: Baseline and 1 year after screening
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 530G Insulin Pump
Number analyzed (Participants) | 3
percentage | 0.37 (0.47)

3. Secondary Outcome: Mean Change in A1C From Baseline to 1 Year, Stratified by Different A1c Subgroups
Description: Mean change in A1C from baseline to 1 year, stratified by different A1c subgroups: A1c 7% to 9%. Among the 132 subjects with both baseline and end of study A1c, 97 had A1c 7% to 9%
Time Frame: Baseline and 1 year after screening
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 530G Insulin Pump
Number analyzed (Participants) | 97
percentage | 0.34 (0.73)

4. Secondary Outcome: Mean Change in A1C From Baseline to 1 Year, Stratified by Different A1c Subgroups
Description: Mean change in A1C from baseline to 1 year, stratified by different A1c subgroups: A1c > 9%. Among the 132 subjects with both baseline and end of study A1c, 32 had A1c > 9%
Time Frame: Baseline and 1 year after screening
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 530G Insulin Pump
Number analyzed (Participants) | 32
percentage | -0.02 (1.27)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 530G Insulin Pump
All-Cause Mortality (participants affected / at risk) | 0/194
Serious Adverse Events (participants affected / at risk) | 4/194
Other Adverse Events (participants affected / at risk) | 121/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 530G Insulin Pump (N=194)
Severe Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Dabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (2)
Second Degree Burns to lower distal extremeties (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 530G Insulin Pump (N=194)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Body dysmorphic disorder (Psychiatric disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Chest pain (General disorders) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear infection (Infections and infestations) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Encephalitis viral (Infections and infestations) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fear of injection (Psychiatric disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (6)
Gastroenteritis viral (Infections and infestations) | 4 (4)
Gastrointestinal viral infection (Infections and infestations) | 2 (2)
Giardia test positive (Investigations) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (2)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3)
Headache (Nervous system disorders) | 6 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 28 (44)
Hypersensitivity (Immune system disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4)
Influenza (Infections and infestations) | 5 (6)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Ketonuria (Renal and urinary disorders) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Medical device discomfort (General disorders) | 1 (1)
Medical device pain (General disorders) | 8 (9)
Medical device site reaction (General disorders) | 17 (23)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Mononucleosis syndrome (Infections and infestations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Onychomycosis (Infections and infestations) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Otitis media (Infections and infestations) | 3 (4)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (3)
Pharyngitis streptococcal (Infections and infestations) | 8 (11)
Pneumonia (Infections and infestations) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 10 (10)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 5 (6)
Skin infection (Infections and infestations) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 20 (28)
Syncope (Nervous system disorders) | 3 (3)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2)
Tuberculin test positive (Investigations) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 18 (22)
Urinary tract infection (Infections and infestations) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1)
Viral infection (Infections and infestations) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-08-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT02120794/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT02120794/SAP_001.pdf